CLINICAL TRIAL: NCT04687150
Title: Fecal Microbiota Transplantation in Newly Diagnosed Ulcerative Colitis Patients
Brief Title: Fecal Microbiota Transplantation and Newly Diagnosed Ulcerative Colitis (UC)
Acronym: FinUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other); Päijänne Tavastia Central Hospital (Other)
Responsible Party: Principal Investigator, Kimmo Salminen, MD, PhD, Specialist in Gastroenterology, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T298/2020
Record Dates: First submitted 2020-11-30; First posted 2020-12-29 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled pilot study. Accrued participants were randomized 1:1 using a computer generated randomization algorithm (www.random.org).
Who Masked: Participant, Care Provider, Investigator
Masking Description: e
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Active Comparator): The study group with newly diagnosed active ulcerative colitis receive an FMT via colonoscopy from a tested general donor, frozen and thawed from a fecal bank at week 0 and at week 4 as an enema at the study nurse´s visit
  Interventions: Other: Fecal microbiota transplantation
- The control group (Placebo Comparator): The control group will be given colored water at same timepoints
  Interventions: Other: Colored water

INTERVENTIONS:
Other: Fecal microbiota transplantation — Fecal microbiota transplantation from a tested general donor, frozen and thawed from a fecal bank
  Arms: The study group
Other: Colored water — Colored water (placebo)
  Arms: The control group

SUMMARY:
In this FinUC study we are trying to find out the efficacy and safety of the Fecal microbiota transplantation (FMT) in newly diagnosed active ulcerative colitis patients. The study group with newly diagnosed active ulcerative colitis receive an FMT via colonoscopy from a tested general donor, frozen and thawed from a fecal bank at week 0 and at week 4 as an enema at the study nurse´s visit. The control group will be given colored water. The main aim of the FinUC study is to determine how the FMT change of the gut microbiota composition in newly diagnosed active ulcerative colitis patients. The other aim is to determine efficacy and mechanisms of fecal microbiota transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Active newly diagnosed colitis (Mayo score <11)
* Signed informed consent

Exclusion Criteria:

* Fulminant severe colitis (Mayo score 11-12 or Truelove and Witts criteria)
* Gastrointestinal infection
* Pregnancy
* Antibiotic therapy at the baseline
* On-going probiotic medication
* Unable to provide signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Modified gut microbiota composition | at week 12
  Increased species richness and alfa-diversity

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo K Salminen, MD,PhD, Study Director — Head of the section
Locations (1):
- Kimmo Salminen, Turku, Finland

IPD SHARING:
Plan to Share IPD: No